CLINICAL TRIAL: NCT06703840
Title: A Phase 2a, Randomised, Double-blind, Parallel and Placebo-controlled Trial Investigating Safety and Efficacy of LIB-01 in Treatment of Erectile Dysfunction
Brief Title: Phase 2a Trial to Investigate the Efficacy of LIB-01 in Treatment of Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dicot AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCT4564
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): LIB-01 Placebo, oral suspension
  Interventions: Drug: LIB-01 Placebo
- LIB-01 10 mg (Experimental): LIB-01 10 mg, oral suspension
  Interventions: Drug: LIB-01
- LIB-01 25 mg (Experimental): LIB-01 25 mg, oral suspension
  Interventions: Drug: LIB-01
- LIB-01 50 mg (Experimental): LIB-01 50 mg, oral suspension
  Interventions: Drug: LIB-01

INTERVENTIONS:
Drug: LIB-01 — LIB-01 oral suspension
  Arms: LIB-01 10 mg; LIB-01 25 mg; LIB-01 50 mg
Drug: LIB-01 Placebo — LIB-01 Placebo oral suspension
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the drug LIB-01 works to treat erectile dysfunction in male adults. It will also learn about the safety of the drug LIB-01. The main questions it aims to answer are:

* Does the drug LIB-01 improve erectile function in males with erectile dysfunction?
* What medical problems do participants have when taking the drug LIB-01? Researchers will compare the drug LIB-01 to a placebo (a look-alike substance that contains no drug) to see if the drug LIB-01 works to treat erectile dysfunction.

Participants will:

* Take the drug LIB-01 or a placebo every day for 3 days
* Visit the clinic every week for 4 weeks, and at 8 weeks, for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any trial specific procedures.
2. Male participant aged 25 to 65 years, inclusive, at the screening visit.
3. In a stable heterosexual relationship for at least 6 months prior to the screening visit.
4. Total score of 11-25 on questions 1-5 and 15 on the EF domain of the IIEF questionnaire.
5. Highly motivated to obtain treatment for ED.
6. Willing to abstain from unprotected sex and use condom to prevent drug exposure of a partner and pregnancy from first dose until the end-of-trial. In addition, refrain from donating sperm from the date of dosing until 3 months after (last) dosing with the IMP. Any female partner of child-bearing potential of a non-vasectomised trial participant must use contraceptive methods with a failure rate of < 1% to prevent pregnancy until the end-of-trial visit.
7. Understands the trial requirements.

Exclusion Criteria:

1. History of any clinically significant disease or disorder, including psychiatric disorder, which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or influence the results or the participant's ability to participate in the trial.
2. Type 1 diabetes.
3. Haemoglobin A1c (HbA1c) ≥48 mmol/L (6.5%).
4. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
5. Malignancy within the past 5 years, with the exception of in situ removal of basal cell carcinoma.
6. Any planned major surgery within the duration of the trial.
7. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to LIB-01 API.
8. History of priapism, or increased risk due to underlying illness, including but not limited to hemoglobinopathies such as sickle cell anaemia or thalassemia.
9. History of glaucoma.
10. History of Non-Arteritic Anterior Ischemic Optic Neuropathy (NAION).
11. History of prostatectomy.
12. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
13. Presence or history of drug abuse, as judged by the Investigator.
14. History of, or current use of anabolic steroids, as judged by the Investigator.
15. Bleeding deficiencies or ongoing anticoagulant therapy that would put the participant at risk, as judged by the investigator.
16. Uncontrolled cardiac disease within 6 months of screening, including but not limited to uncontrolled hypertension; unstable angina; myocardial infarction or cerebrovascular accident.
17. Use of nitrate medications within 14 days prior to the screening visit.
18. Use of any drug with narrow therapeutic index or drugs that are sensitive substrates, strong inducers or strong inhibitors to CYP3A4 as well as substrates and inhibitors of OATP1B1 or sensitive to substrates to CYP2B6 in accordance with the list provided (see Section 9.6.2.1).
19. Use of oral, injectable, intra-urethral, or topical pro-erectile drugs or supplements, including but not limited to PDE5-Is or prostaglandin E1, or use of devices for ED treatment, within 14 days prior to screening.
20. Primary hypoactive sexual desire.
21. Presence of penile anatomical abnormalities, such as penile fibrosis or Peyronie's disease, which would cause significantly impaired sexual performance, as judged by the Investigator.
22. Insufficient therapeutic effect when using PDE5-Is.
23. History of, or ongoing antiandrogen treatment.
24. Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis B and C antibodies and/or human immunodeficiency virus (HIV).
25. Abnormal vital signs, laboratory test value or ECG of clinical significance, as judged by the Investigator.
26. Moderate to severe renal impairment with an eGFR (creatinine) ≤60 mL/min (revised Malmö-Lund equation).
27. Moderate to severe hepatic impairment at the time of the screening visit, as judged by the Investigator.
28. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the last three months prior to the screening visit.
29. Planned treatment or treatment with another investigational therapy (i.e., small molecule or biologic) within 3 months prior to the screening visit.
30. Involvement in the planning, and/or conduct of the trial.
31. The Investigator considers the participant unlikely to comply with trial procedures, restrictions and requirements.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-07-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of LIB-01 in the treatment of erectile dysfunction (ED). | 4 weeks
  Change from baseline in total score on the erectile function (EF) domain of the patient questionnaire International Index of Erectile Function (IIEF-EF) at week 4.

SECONDARY OUTCOMES:
To evaluate the efficacy of LIB-01 in improving erectile function (ability to penetrate) during sexual intercourse. | 8 weeks
  Percentage of successful attempts by the Sexual Encounter Profile (SEP) question 2 throughout the trial period.
To evaluate the efficacy of LIB-01 in improving erectile function (maintained for completion) during sexual intercourse. | 8 weeks
  Percentage of successful attempts by the Sexual Encounter Profile (SEP) question 3 throughout the trial period.
To evaluate the efficacy of LIB-01 in improving erections. | 8 weeks
  Percentage of improved erections by the Global Assessment Question (GAQ) at week 4 and week 8.
To evaluate the incidence of treatment-emergent adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) following oral dosing of LIB-01 | 8 weeks
  Frequency, seriousness and intensity of adverse events (AEs). Adverse events will be graded from 1-5 by the Common Terminology Criteria for Adverse Events (CTCAE):
  Grade 1, Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2, Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL).
  Grade 3, Severe or medically significant but not immediately life-threatening; hospitalisation or prolongation of hospitalisation indicated; disabling; limiting self- care ADL.
  Grade 4, Life-threatening consequences: urgent intervention indicated. Grade 5, Death related to AE.
To evaluate changes in vital signs (blood pressure), following oral dosing of LIB-01. | 8 weeks
  Clinically significant changes in blood pressure.
To evaluate changes in vital signs (pulse), following oral dosing of LIB-01. | 8 weeks
  Clinically significant changes in pulse.
To evaluate changes in vital signs (respiratory rate), following oral dosing of LIB-01. | 8 weeks
  Clinically significant changes in respiratory rate.
To evaluate changes in vital signs (body temperature), following oral dosing of LIB-01. | 8 weeks
  Clinically significant changes in vital body temperature.
To evaluate changes in ECG parameters (resting heart rate [HR]), following oral dosing of LIB-01. | 8 weeks
  Clinically significant changes in resting heart rate (HR).
To evaluate changes in ECG parameters (PQ/PR), following oral dosing of LIB-01. | 8 weeks
  Clinically significant changes in PQ/PR interval.
To evaluate changes in ECG parameters (QRS), following oral dosing of LIB-01. | 8 weeks
  Clinically significant changes in QRS interval.
To evaluate changes in ECG parameters (QT), following oral dosing of LIB-01. | 8 weeks
  Clinically significant changes in QT interval.
To evaluate changes in ECG parameters (QTcF [corrected QT interval by Fredericia]), following oral dosing of LIB-01. | 8 weeks
  Clinically significant changes in QTcF interval.

CONTACTS AND LOCATIONS:
Locations (6):
- Herlev Hospital, Herlev, Herlev, Denmark
- Clinical Trial Consultants, Groningen, Provincie Groningen, Netherlands
- Sweden (4):
  - Clinical Trial Consultants, Mölndal, Göteborg
  - Clinical Trial Consultants, Linköping, Linköping
  - Clinical Trial Consultants, Solna, Stockholm County
  - Clinical Trial Consultants, Uppsala, Uppsala County

IPD SHARING:
Plan to Share IPD: Yes